CLINICAL TRIAL: NCT06882083
Title: The Effect of Ultrasound-Guided Bilateral Single-Shot Paravertebral Block on Recovery After Coronary Artery Bypass Graft Surgery
Brief Title: The Effect of Paravertebral Block on Recovery After CABG Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Associate Professor, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ADYU-ANS-NY-009
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Bypass Surgery; Paravertebral Block
Keywords: Paravertebral block; Coronary artery bypass surgery; Quality of recovery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers who performed the blocks did not participate in the outcome assessments, and similarly, the researcher evaluating the outcomes was not involved in the paravertebral block procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): No intervention planned for control group. Patients in the control group will receive a standard analgesia protocol.
- Block group (Experimental): USG guided single-shot paravertebral block planned for block group
  Interventions: Procedure: paravertebral block

INTERVENTIONS:
Procedure: paravertebral block — A single-dose bilateral paravertebral block will be administered under ultrasound guidance before the induction of general anesthesia. The block will be performed at an appropriate thoracic level using 20 mL of 0.25% bupivacaine as the local anesthetic.
  Arms: Block group

SUMMARY:
The study aims to evaluate the analgesic efficacy of paravertebral block, mobilization speed, respiratory functions, and complication rates in patients who have undergone cardiac surgery and are monitored in the intensive care unit during the postoperative period.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of a single-dose bilateral paravertebral block administered under ultrasound guidance on the recovery process after cardiac surgery. Effective management of postoperative pain in cardiac surgeries is crucial for enhancing patient comfort, reducing complications, and facilitating rapid recovery. Paravertebral block can be utilized as an effective method for pain management following cardiac surgeries. This technique provides extensive analgesic coverage in the thoracic region while reducing opioid consumption and its associated side effects. Additionally, it supports the preservation of respiratory functions, facilitates early mobilization, and may reduce postoperative complications. When performed under ultrasound guidance, the accuracy and efficacy of the block are enhanced, making it a safe analgesic option in cardiac surgeries. Studies have demonstrated that paravertebral block increases patient satisfaction and contributes positively to the recovery process. Therefore, it is a viable approach for postoperative pain management in cardiac surgery.

This study will be conducted with a prospective, randomized, and controlled design. Patients will be assigned to two groups using a sealed-envelope method: the paravertebral block group and the control group. Patients in the paravertebral block group will receive a single-dose bilateral paravertebral block under ultrasound guidance before the induction of general anesthesia. The block will be performed at an appropriate thoracic level using 20 mL of 0.25% bupivacaine as the local anesthetic. Patients in the control group will receive a standard analgesia protocol.

All patients will be monitored in the intensive care unit during the postoperative period, and the following parameters will be assessed: pain scores using the visual analog scale (VAS), total opioid consumption, extubation times, intensive care unit length of stay, Quality of Recovery-15 (QoR-15) score, and postoperative complications. Data will be collected during the preoperative assessment and throughout the first 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older scheduled for elective coronary artery bypass graft surgery with median sternotomy

Exclusion Criteria:

* Contraindications to neuroaxial block ( coagulopathy, infection at the injection site, allergy to local anesthetics..)
* Emergency surgeries
* severe back deformities
* Chronic pain
* refusal to participate
* CABG without sternotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery -15 (QoR-15) score | Postoperative 24th hours
  The QoR-15 is a clinically acceptable and feasible patient-centred outcome measure after surgery. The score demonstrated good validity, reliability and responsiveness. The score ranges from 0 to 150. O refers to the worst recovery and 150 refers to best recovery.

SECONDARY OUTCOMES:
Visual Analog scale (VAS) score | Postoperative 2nd, 4th, 6th, 12th and 24th hours
  The Visual Analog Scale (VAS) score is a pain assessment tool. The score ranges from 0 to 10, with 0 indicating no pain and 10 indicating the worst pain ever experienced
Opioid consumption | Postoperative 24th hours
  Total opioid consumption in first postoperative day will be recorded
Extubation time | Time frame from the end of the surgery to extubation
  Time frame from the end of the surgery to extubation will be recorded

IPD SHARING:
Plan to Share IPD: Undecided